CLINICAL TRIAL: NCT01545752
Title: Comparing Interactive and Non-interactive CD-based Method in Teaching Medical Terminology
Brief Title: Comparing Interactive and Non-interactive CD-based Method
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nazila zarghi, principal investigator, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CD-based education
Record Dates: First submitted 2012-02-22; First posted 2012-03-07 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-03

CONDITIONS: Interactive CD-based Education
Keywords: elearning; CD-based education
MeSH Terms: interventions — CD-I

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- coventional group (No Intervention): Teaching just by book
- non-interactive CD (Experimental): Teaching book with non-interactive CD
  Interventions: Other: teaching by non-interactive CD
- interactive CD (Experimental): Teaching book with interactive CD
  Interventions: Other: Interactive CD

INTERVENTIONS:
Other: teaching by non-interactive CD — teaching book with non-interactive CD
  Arms: non-interactive CD
Other: Interactive CD — Teaching book with interactive CD
  Arms: interactive CD

SUMMARY:
Using different methods of electronic learning has been increasingly developed by emerging electronic educational technologies. They could apply on the net, CDs, Mobile, etc in different usage alternatives: interactive and non-interactive both in online and off-line approaches. In this educational trial, the interactive and non-interactive CD-based method for teaching medical terminology to nursing students of MUMS school of nursing and Midwifery during 2009-2012 was compared.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students studying in MUMS school of nursing and passing Medical Terminology

Exclusion Criteria:

* any other discipline,
* students of other schools

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
students' mean Scores | up to three years
  the outcome mesures will be completed up to 6 months